CLINICAL TRIAL: NCT03030391
Title: Evaluation of a Novel Positron Emission Tomography (PET) Radiotracer to Image Phosphodiesterase-4B (PDE4B)
Brief Title: Novel Positron Emission Tomography (PET) Radiotracer to Image Phosphodiesterase-4B (PDE4B)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 170041; 17-M-0041
Record Dates: First submitted 2017-01-24; First posted 2017-01-25 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2018-03-16

CONDITIONS: Healthy
Keywords: Camp; Radiation Absorbed Dose; Compartmental Analysis
MeSH Terms: conditions — Muscle Cramp

INTERVENTIONS:
Other: PET
Other: MRI

SUMMARY:
Background:

The new drug 18F-PF-06445974 has a little radioactivity. This can be seen by a positron emission tomography (PET) scan. The drug helps researchers see a protein, PDE4B, in the brain. Looking at PDE4B in the living brain might show how it is involved in psychiatric and neurological disorders. One part of the study will look at how the study drug is distributed in the brain. Another part will study how brain measures vary.

Objectives:

To measure the protein PDE4B in the brain. To test how a new radioactive chemical, 18F-PF-06445974, is distributed in the body.

Eligibility:

Healthy adults ages 18 and older

Design:

Participants will have 1-3 visits over a year. Each will be 2-5 hours.

Women will have a pregnancy test each time.

DETAILED DESCRIPTION:
Objective:

Phosphodiesterase type 4 (PDE4) terminates signal transduction of guanine nucleotidebinding proteins (G-protein)-coupled receptors by metabolizing the second messenger 3 <=,5 <=- cyclic adenosine monophosphate (cAMP). PDE4 is selective to cAMP over cyclic guanosine monophosphate. PDE4 has four isozymes A, B, C, and D and basic studies indicate that type B (PDE4B) plays a key role in cognitive function and neuroinflammation. Thus, PDE4B inhibitors would be expected to improve cognitive function and have anti-inflammatory effects. Pfizer has developed a new PET ligand, 18F-PF-06445974, to selectively image PDE4B; the ligand has shown promising results in non-human primates.

This protocol covers four phases:

1. Phase 1: whole body imaging of one subject with a low injection activity of 2 mCi to confirm that no organ has prominently high uptake of 18F-PF-06445974;
2. Phase 2: kinetic brain imaging with up to 5 mCi injection to quantify PDE4B in brain relative to concurrent measurement of the parent radioligand in arterial plasma;
3. Phase 3: if 18F-PF-06445974 is successful in Phase 2 in the first couple of subjects, we will estimate the radiation-absorbed doses by performing whole body imaging with 5 mCi injection;
4. Phase 4: test-retest analysis of brain binding relative to concurrent measurement of the parent radioligand in arterial plasma (5 mCi per scan).

Study Population:

Healthy adult female and male volunteers (n=22, ages 18 or older) will undergo brain imaging. An additional eight healthy volunteers will undergo whole body dosimetry analysis, for a total of 30 healthy volunteers.

Design:

For quantification of 18F-PF-06445974, 22 healthy controls will undergo brain PET imaging using 18F-PF-06445974 and an arterial line. Some of them will have a test-retest scan. Eight additional subjects will have a whole body PET scan for dosimetry. For dosimetry, no arterial line will be used.

Outcome Measures:

To assess quantitation of PDE4B with 18F-PF-06445974, we will primarily use two outcome measures, namely the identifiability and time stability of distribution volume (VT) calculated with compartmental modeling. In the test-retest study, we will calculate the retest

variability. We will assess whole-body biodistribution and dosimetry of 18F-PF-06445974 by calculating doses to organs and effective dose to the body.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18 or older.
* Able to give written informed consent.
* Medically and psychiatrically healthy.
* Enrolled in 01-M-0254 The Evaluation of Participants with Mood and Anxiety Disorders and Healthy Volunteers (PI: Dr. Carlos Zarate).

EXCLUSION CRITERIA:

* Any current Axis I diagnosis.
* Clinically significant laboratory abnormalities
* Positive HIV test.
* Unable to have an MRI scan.
* History of neurologic illness or injury with the potential to affect study data interpretation.
* Recent exposure to radiation related to research (i.e. PET from other research) that, when combined with this study, would be above the allowable limits.
* Inability to lie flat on camera bed for at least two hours.
* Pregnancy or breastfeeding.
* Current substance use disorder based on DSM-5.
* Current use of psychiatric medications.
* NIMH employees/staff and their immediate family members will be excluded from the study per NIMH policy.

Exclusion criteria for the dosimetry subjects are the same as reported above, with the exception of MRI contraindications, because an MRI will not be performed in these subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-01-10; Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
Quantification of 18F-PF-06445974 binding in brain | 2 hours

SECONDARY OUTCOMES:
Biodistribution of 18F-PF-06445974 in the body. | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Fujita, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States